CLINICAL TRIAL: NCT01799603
Title: A Single-dose, Open-label, Randomized, Two-way Crossover Study to Assess the Effect of Food on the Pharmacokinetics of TMC435 in Japanese Healthy Adult Male Subjects
Brief Title: A Pharmacokinetic Study to Assess the Effect of Food in Healthy Male Participants Receiving TMC435
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100854; TMC435HPC1007
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: Healthy; TMC435; G008
MeSH Terms: interventions — Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TMC435 in fasted then fed condition (Experimental): Participants under fasting condition will be administered with TMC435, 100 milligram (mg) as oral capsule on Day 1 of first treatment period and then will be administered with TMC435, 100 mg oral capsule on Day 1 under fed condition of second treatment period (after washout period of 9 days, between the two treatment periods).
  Interventions: Drug: TMC435
- TMC435 in fed then fasted condition (Experimental): Participants under fed condition will be administered with TMC435, 100 milligram (mg) as oral capsule on Day 1 of first treatment period and then will be administered with TMC435, 100 mg oral capsule on Day 1 under fasting condition of second treatment period (after washout period of 9 days, between the two treatment periods).
  Interventions: Drug: TMC435

INTERVENTIONS:
Drug: TMC435 — TMC435, 100 milligram oral capsule will be administered on Day 1 of each treatment period, separated by washout period of 9 days.
  Other Names: G008

SUMMARY:
The purpose of this study is to investigate the effect of food on the pharmacokinetics (explores what the body does to the drug) and safety of TMC435 in Japanese healthy adult male participants.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-center, 2-way crossover (method used to switch participants from one treatment arm to another in a clinical trial) and randomized (the study drug is assigned by chance) study to assess the effect of food on the pharmacokinetics of TMC435 after a single dose in Japanese healthy adult male participants. The study duration will be of 44 days per participant, which is divided into 3 parts: Screening (from Day -28 to Day -2); Treatment (consists of 2 treatment periods of 5 days each [that is, Day -1 to 4, in-patient period], wherein all participants will receive TMC435 in the respective period, and the period will be separated by washout period of 9 days); and Follow-up (on Day 7 of Period 2). Participants will keep upright position from the time of study drug administration until 4 hours after study drug administration. Participants will not be allowed to ingest meal until 4 hours post-dose. Participants will have standardized lunch and dinner at 4 hours and 10 hours post-dose, respectively. Drinking water will not be allowed from 1 hour before the administration up to 1 hour after administration except for the water served with the study drug and meal. Pharmacokinetics will be assessed in blood samples which will be collected up to 72 hours after administration of study drug. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Be a Japanese man aged 20 to 40 years, inclusive at the day of informed consent being signed
* Must agree to use an adequate contraception method (for example, double-barrier method) as deemed appropriate by the Investigators during the study and for 3 months after receiving the last dose of study drug
* Body mass index (BMI) between 18.5 and 25.0 kilogram per square meter (kg/m^2) and body weight not less than 50 kilogram
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic
* Non-smoker or participant who has quitted any tobacco or nicotine containing products more than one year prior to screening

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to), cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the Investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Use of any prescription or non-prescription medication (including vitamins and supplements) within 14 days before the administration on Day 1 of treatment Period 1
* History of drug or alcohol abuse within the past 5 years and positive test for drugs of abuse, such as cannabinoids, opiates, cocaine, amphetamines, benzodiazepines or barbiturates and serum alcohol test
* Known allergy to the study drug or any of the excipients of the formulation
* Participated in another clinical study and received another study drugs administration or used an experimental medical device within 120 days or within a period less than 10 times the drug's half life, whichever is longer, before Day 1 of the first treatment period

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (C[max]) | -3 hours (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose on Day 1
  The C(max) is the maximum plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[infinity]) | -3 hours (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose on Day 1
  The AUC (infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC (last) and C (last)/lambda (z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C (last) is the last observed quantifiable concentration; and lambda (z) is elimination rate constant.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Toshima City, Japan